CLINICAL TRIAL: NCT05291182
Title: A First-in-human, Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Anti-tumor Activity of SY-4835 Tablets in Patients With Advanced Solid Tumor
Brief Title: A Phase I Study of SY-4835 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shouyao Holdings (Beijing) Co. LTD (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SY-4835-1
Record Dates: First submitted 2022-03-02; First posted 2022-03-22 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-04

CONDITIONS: Advanced Solid Tumor
Keywords: SY-4835; WEE1; Advanced solid tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose-escalation (Experimental): The study is conducted to evaluate the safety, tolerability, pharmacokinetics (PK) and anti-tumor activity of SY-4835.
  Interventions: Drug: SY-4835

INTERVENTIONS:
Drug: SY-4835 — WEE1 inhibitor
  Other Names: SY-4835 tablets

SUMMARY:
This is a phase 1, open-label, single-arm, first-in-human study to evaluate the safety, tolerability, pharmacokinetics (PK) and anti-tumor activity of SY-4835 administered orally in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study is a first-in-human phase I study of SY-4835, a potent WEE1 inhibitor, in patients with advanced solid tumor. Dose-escalation study is conducted to evaluate primary endpoints and secondary endpoints including the maximum tolerated dose (MTD), Dose-limiting toxicity (DLT), pharmacokinetics (PK) parameters and recommended phase II dose (RP2D), and the safety, tolerability and pharmacokinetics (PK) profiles of SY-4835 are characterized in this study.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion in this study, patients must fulfil the following criteria:

  1. Must understand andvoluntarily sign the informed consent form, willing to follow and able to complete all study procedures.
  2. Male or female (age of 18~75 years old ).
  3. Eastern Collaboration Oncology Group (ECOG) performance status (PS) scored of 0-1.
  4. Estimated life expectancy ≥3 months.
  5. Histological or cytological confirmation of a advanced solid tumor, that failed to respond to standard therapy, progressed despite standard therapy, or for which standard therapy does not exist.
  6. At least 1 measureable lesion for solid tumors assessed using RECIST 1.1.
  7. Patients must have adequate organ function as defined below (no supportive treatment for the following parameters within 7 days prior to testing):

     Liver function:

     Patients without hepatic metastasis, aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 3 times institutional upper limit of normal (ULN), total bilirubin (TBIL) ≤ 1.5 times ULN; Patients with hepatic metastasis, AST, ALT ≤ 5 times ULN, TBIL ≤ 1.5 times ULN; Patients with hepatoma carcinoma, AST and ALT ≤ 5 times ULN, TBIL ≤ 2.5 times ULN.

     Bone marrow function:

     Absolute neutrophil count (ANC) ≥ 1.5×10^9/L; Platelets (PLT) count ≥ 75×10^9/L; Hemoglobin (HB) ≥ 80 g/L.

     Renal function:

     Creatinine clearance ≥ 45 mL/min or serum creatinine ≤ 1.5 times ULN.

     Coagulation function:

     Activated partial thromboplastin time (APTT) ≤ 1.5×ULN; International Normalized ratio (INR) ≤ 1.5×ULN.
  8. Women of childbearing age performed a serum pregnancy test within 7 days before the initiation of treatment, and agreed to adopt a reliable and effective contraceptive method during the trial and within 90 days after the final administration of the study drug.

Exclusion Criteria:

* Patients must not enrol in this study if any of the following exclusion criteria are fulfilled:

  1. Have received chemotherapy, radiotherapy, biotherapy, endocrine therapy, immunotherapy and other anti-tumor therapy within 3 weeks prior to the first use of the study drug, except for the following:

     Nitrosourea or mitomycin C were used within 6 weeks prior to the first use of the study drug; Oral fluorouracil and small molecule targeted drugs were used within 2 weeks or within 5 half-lives prior to the first use of the study; Chinese medicines were used within 2 weeks prior to the first use of the study drug.
  2. Have received an unmarketed clinical investigational drug or treatment within 4 weeks prior to the first use of the study drug.
  3. Had major organ surgery (excluding needle biopsy) or had significant traumatism within 4 weeks prior to the first use of study drug.
  4. History of any WEE1 inhibitor treatment.
  5. With the exception of alopecia and ≤ Grade 2 peripheral neuropathy, any unresolved toxicities from prior treatment ≤ Grade 1 according to the Common Terminology Criteria for Adverse Events (CTCAE) at the time of starting study treatment.
  6. Evidence of central nervous system (CNS) metastases accompanied with clinical symptoms, or other evidence of uncontrolled CNS metastases judged by investigators that the patient should not participate in the study.
  7. Patients have serous effusion (such as pleural effusion, peritoneal effusion, pericardial effusion, etc.) with clinical symptoms, effusions will still increase after 2 weeks of conservative treatment (excluding drainage).
  8. Patients with active uncontrolled systemic bacterial, viral, or fungal infection despite optimal treatment.
  9. Active hepatitis B (HBsAg-positive and HBV-DNA ≥ 2000 IU/ mL), Hepatitis C virus infection (HCVAb-positive and HCV-RNA ≥ 1000 IU/ml); Human immunodeficiency virus antibody (HIV Ab) positive; Active syphilis.
  10. Have serious cardiovascular and cerebrovascular diseases, including but not limited to:

      Severe arrhythmias or abnormal cardiac conduction, such as ventricular arrhythmias requiring clinical intervention, degree ii-iii atrioventricular block, etc; Mean resting corrected QT interval (QTcF) > 470 msec obtained from 3 electrocardiograms (ECGs); Had acute coronary syndrome, congestive heart failure, aortic dissection, or other grade 3 or higher cardio-cerebrovascular events within 6 months prior to the first use of study drug; Heart failure (New York Heart Association, NYHA) class ≥ II or left ventricular ejection fraction (LVEF) < 40 %; Hypertension remains uncontrolled after aggressive antihypertensive therapy. Uncontrolled hypertension was defined as systolic blood pressure > 185 mmHg and/or diastolic blood pressure > 110 mmHg measured on 3 repetitions at least 10 minutes apart.
  11. Prescription or non-prescription drugs known as moderate to strong inhibitors / inducers of CYP3A4 and CYP2D6 within 7 days prior to the first dose of study treatment.
  12. Patients with alcohol and/or drug dependence.
  13. Women who are breastfeeding.
  14. Patients suffering from conditions which are likely to adversely affect gastrointestinal motility.
  15. Patients with malignancies other than tumors treated in this study (except: malignancies that are cured and have not recurred within 3 years prior to study entry; completely resected basal cell and squamous cell skin cancer; completely resected carcinoma in situ of any type).
  16. The investigator considers that the subject has a history of other serious systemic diseases or other reasons and is not suitable to participate in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-28 (Actual); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-12-28 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AE), serious adverse events (SAEs), suspected unexpected serious adverse reaction (SUSAR), physical examination, etc. (CTCAE 5.0 standard) | Up to 24 months
  Characterization of the safety and tolerability
Tolerability: Ratio of Dose reductions or interruptions | Up to 24 months
  Characterization of the safety and tolerability
Incidence rate of dose limiting toxicities (DLTs) | cycle 1 (each cycle is 21 days)
  Maximum Tolerated Dose(s) (MTD(s)) and recommended phase 2 dose (RP2D(s))

SECONDARY OUTCOMES:
Pharmacokinetics (Cmax) for SY-4835 | Cycle 1 (each cycle is 21 days)
  Defined as maximum observed plasma concentration
Pharmacokinetics (Tmax) for SY-4835 | Cycle 1 (each cycle is 21 days)
  Defined as time to maximum plasma concentration
Pharmacokinetics (AUC0-t) for SY-4835 | Cycle 1 (each cycle is 21 days)
  Defined as area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration
Pharmacokinetics (t½) for SY-4835 | Cycle 1 (each cycle is 21 days)
  Defined as the apparent plasma terminal phase disposition half-life
Overall Response Rate (ORR) as assessed by RECIST 1.1 criteria | Up to 24 months
  Preliminary measure of anti-tumor activity of SY-4835
Progression Free Survival (PFS) | Up to 24 months
  Preliminary measure of anti-tumor activity of SY-4835
Disease control rate (DCR) | Up to 24 months
  Preliminary measure of anti-tumor activity of SY-4835
Duration of response (DOR) | Up to 24 months
  Preliminary measure of anti-tumor activity of SY-4835

CONTACTS AND LOCATIONS:
Overall Officials: Yinghui Sun, PhD, Study Director — Shouyao Holdings (Beijing) Co. LTD
Locations (1):
- Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No